CLINICAL TRIAL: NCT00670917
Title: A Randomized Controlled Trial Assessing the Effect of Magnetic Acupressure in Reducing Pain in Cancer Patients Undergoing Bone Marrow Aspiration and Biopsy
Brief Title: Magnetic Acupressure in Reducing Pain in Cancer Patients Undergoing Bone Marrow Aspiration and Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: J07103; P30CA006973 (NIH); CDR0000594676; NA_00013389 (Other: JHM IRB)
Record Dates: First submitted 2008-05-01; First posted 2008-05-02 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Hematopoietic/Lymphoid Cancer; Pain
Keywords: pain; hematopoietic/lymphoid cancer
MeSH Terms: conditions — Hematologic Neoplasms; Pain | interventions — Acupressure; Biopsy; Analgesia

ARMS (2):
- L14 acupoint (Active Comparator)
  Interventions: Other: questionnaire administration; Procedure: acupressure therapy; Procedure: biopsy; Procedure: bone marrow aspiration; Procedure: pain therapy
- Sham Point (Sham Comparator)
  Interventions: Other: questionnaire administration; Procedure: acupressure therapy; Procedure: biopsy; Procedure: bone marrow aspiration; Procedure: pain therapy

INTERVENTIONS:
Other: questionnaire administration
Procedure: acupressure therapy
Procedure: biopsy
Procedure: bone marrow aspiration
Procedure: pain therapy

SUMMARY:
RATIONALE: Acupressure may help relieve pain in cancer patients undergoing bone marrow aspiration and biopsy. It is not yet known whether magnetic acupressure is more effective than sham acupressure in reducing pain in cancer patients undergoing bone marrow aspiration and biopsy.

PURPOSE: This randomized clinical trial is studying magnetic acupressure to see how well it works compared with sham acupressure in reducing pain in cancer patients undergoing bone marrow aspiration and biopsy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare pain rating in cancer patients undergoing bone marrow aspiration and biopsy (BMAB) treated with magnetic acupressure at bilateral large intestine 4 (LI 4) points vs sham acupressure at bilateral proximal fourth interosseus space of the hand.

Secondary

* To compare the duration of BMAB, patient's rating of the procedure, and patient's willingness to receive acupressure during subsequent BMABs.

OUTLINE: Patients are stratified according to the number of prior bone marrow aspirations and biopsies (BMAB) (0-1 vs ≥ 2) and type of procedure (bone marrow aspiration alone vs BMAB). Patients are randomized to one of two treatment arms.

* Arm I (acupressure): Patients receive acupressure at bilateral large intestine 4 (LI 4) points using Haci Magnetic Acupressure Suction Cups (MASC) during BMAB.
* Arm II (sham acupressure): Patients receive acupressure at bilateral proximal fourth interosseus space of the hand using the same size MASC as in arm I during BMAB.

Patients in both arms also receive analgesic and anxiolytic medications as determined by the acupressure operator and physician.

Patients complete a questionnaire before and after BMAB to assess pain experienced before and during BMAB and their attitude towards the procedure.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer
* Scheduled to undergo a routine bone marrow aspiration with or without biopsy

  * No requirement for conscious sedation during the procedure

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior acupuncture or acupressure
* No prior participation in this study

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2008-05-07 (Actual); Primary Completion 2010-01-19 (Actual); Study Completion 2010-01-19 (Actual)

PRIMARY OUTCOMES:
Pain scores before and during bone marrow aspiration and biopsy (BMAB) as measured by a patient-reported 11-point visual analogue pain scale | 12 hours

SECONDARY OUTCOMES:
Clinical benefit response as measured by duration of BMAB, patient's rating of the procedure, and patient's willingness to receive acupressure during subsequent BMAB | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A. Grossman, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States